CLINICAL TRIAL: NCT06737380
Title: A Phase I, Open-Label Study to Evaluate the Safety and Tolerability of Subcutaneous Administration of Umbilical Cord Derived - Mesenchymal Stromal Cell Therapy in Addition to Standard of Care as A Treatment For Active Systemic Lupus Erythematosus
Brief Title: UC-MSC Cell Therapy Study for Systemic Lupus Erythematosus (SLE) Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LiveKidney.Bio (Industry)
Collaborators: Medical University of South Carolina (Other); Galilee CBR (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LK-23-01
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: SLE; Lupus; Systemic Lupus Erthematosus; Systemic Lupus Erythematosus; Systemic Lupus Erythematosus (SLE)
Keywords: systemic lupus erythematosus; SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Physical Examination; Electrocardiography; Pregnancy Tests; Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UC-MSC therapy (Experimental)
  Interventions: Diagnostic Test: Physical examination; Diagnostic Test: Electrocardiogram; Other: SF-36 questionnaire; Diagnostic Test: Clinical laboratory evaluations - Serology; Diagnostic Test: Clinical laboratory evaluations - Biochemistry; Diagnostic Test: Clinical laboratory evaluations - Hematology; Diagnostic Test: Pregnancy Test; Diagnostic Test: Urinalysis; Diagnostic Test: SLE activity evaluation; Diagnostic Test: SLE biomarker profiling; Diagnostic Test: Cytokines and chemokine profiling; Biological: single dose of UC-MSCs; Other: PROMIS instruments

INTERVENTIONS:
Diagnostic Test: Physical examination — The physical examination will be performed at the Screening visit and at each subsequent study and safety in clinic follow-up visit. The exam will include: measurement of vital signs (heart rate, peripheral arterial blood pressure, respiratory rate, and temperature), weight, height (at Screening visit only), cardiovascular and respiratory systems, abdominal examination, skin evaluation, mouth and eye evaluation, and neurological assessment. Abnormal findings will be recorded in the CRF.
Diagnostic Test: Electrocardiogram — A twelve-lead electrocardiogram (ECG), including corrected QT interval (QTc interval), will be performed in all participants at the Screening visit.
Other: SF-36 questionnaire — Patients will fill out the SF 36 survey, assessing physical and mental health outcomes prior to dosing and/or any other clinical assessments, on visits 1 (baseline), visit 5 (day 14), visit 6 (day 28), visit 11 (day 168) and early termination visit.
Diagnostic Test: Clinical laboratory evaluations - Serology — Serologic testing for HIV, HBV, HCV, TB, and CMV will be performed; HBV and HCV PCR will be done only if serology is positive. Autoimmune tests (ANA, anti-ENA, total IgG, anti-nucleosome) will be done at Day 0 and end of study; ANA only at Screening if no positive ANA or anti-dsDNA in prior 6 months. Inflammatory markers (hs-CRP, ESR) will be tested at Day 0 and end of study. CBC with differential, biochemistry, anti-dsDNA, and complement C3/C4 will be assessed at each scheduled visit.
Diagnostic Test: Clinical laboratory evaluations - Biochemistry — The panel will include analysis of albumin, blood urea nitrogen (BUN), creatinine, glucose, uric acid, calcium, phosphorus, potassium, sodium, lactate dehydrogenase (LDH), total protein, magnesium, alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin and hs-CRP. For biochemistry, 3 mL blood will be collected at each study visit. Results relating to inclusion criteria must be confirmed within 7 days prior to Day 1.
Diagnostic Test: Clinical laboratory evaluations - Hematology — The complete blood count (CBC) will include: hemoglobin, hematocrit, white blood cells (WBCs) with complete manual or automated differential (total neutrophils, lymphocytes, monocytes, eosinophils, basophils; absolute or percentage will be acceptable), red blood cells (RBCs), platelet count. For CBC, 1mL blood will be collected at each study visit.
Diagnostic Test: Pregnancy Test — A serum b-hCG pregnancy test will be performed for women of child-bearing potential at the Screening visit;urine pregnancy tests will be performed for women of child-bearing potential at each study visit noted above, including on Day 0 prior to study treatment.
  Pregnancy tests are not required for women unable to become pregnant for one of the following reasons: Menopause confirmed by healthcare provider, verbally reported by a participant that she has had her uterus or both ovaries or both fallopian tubes removed.
Diagnostic Test: Urinalysis — General urinalysis will include analysis of pH, specific gravity, protein, glucose, ketones, bilirubin, urobilinogen, leukocytes, erythrocytes. In addition samples will be assessed for presence of urinary casts. Spot urine protein/creatinine measure will be done at each visit. If no casts are observed at Screening, then machine assessment of further urinary samples is allowed. For urinalysis, 10mL urine will be collected at each study visit.
Diagnostic Test: SLE activity evaluation — SLE status will be assessed using the Safety of Estrogens in Lupus Erythematosus National Assessment- SLE Disease Activity Index (SLEDAI 2K scale).SLE activity will also be assessed using British Isles Lupus Assessment Group (BILAG), physician global and participant global assessment allowing use of the Systemic Lupus Responder Index (SRI 4) and the BILAG-based Composite Lupus Assessment (BICLA) instruments to assess clinical response.
Diagnostic Test: SLE biomarker profiling — SLE biomarkers will be profiled at the study visit (Day 1) and at every subsequent follow up visit. For this purpose, urine and 10 ml blood will be collected.
  Anti-ENA, Anti-dsDNA antibodies, total serum IgG levels, CBC, C3, C4, anti-nucleosome antibodies, erythrocyte sedimentation rate, CRP, protein/creatinine ratio in spot urine, 24-hour urine protein - Day 1 - Baseline and at end of study visit only; Mononuclear cell changes. This analysis includes lymphocyte subsets and innate immune cell subsets
Diagnostic Test: Cytokines and chemokine profiling — Samples will be analyzed for the following cytokines/chemokines: IFNγ, IL-6, IL-10, IL-18, TNFα, TGFβ1, CXCL10, CCL2, N-GAL, urine endothelin, KIM1. Serum and urine samples will be collected on Days 0, 28, 56, 140, 168, and early termination visit.
Biological: single dose of UC-MSCs — participants will be treated on Baseline Day 1 with a UC-MSCs product administered subcutaneously. Participants will be observed for 2 to 3 hours after end of study treatment and then followed up for safety assessments over the subsequent 6-month period.
Other: PROMIS instruments — PROMIS Fatigue, PROMIS, Depression, PROMIS Pain prior to dosing and/or any other clinical assessments, on visits 1 (baseline, day 0), visit 5 (day 14), visit 6 (day 28), visit 11 (day 168) and early termination visit.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of UC-MSCs in adults with systemic lupus erythematosus (SLE).

The main questions this study aims to answer are:

1. Can UC-MSCs improve kidney function and reduce SLE disease activity?
2. Are UC-MSCs safe and well-tolerated in this patient population?

Participants in this study will:

* Receive UC-MSCs in a single dose in addition to standard of care treatment.
* Provide blood and urine samples for laboratory assessments, including biomarkers and immune profiling (e.g., cytokines, complement proteins, and autoantibodies).
* Attend regular clinic visits for physical exams, disease activity scoring, and imaging tests to monitor kidney health.
* Complete assessments for safety, such as monitoring for adverse events and changes in laboratory values.

This study aims to provide new insights into treatment options for SLE and lupus nephritis, addressing an unmet medical need in this population.

ELIGIBILITY:
Inclusion Criteria

1. Age 18-75 years at the time of screening
2. Diagnosis of systemic lupus erythematosus (SLE), meeting at least 4 of the 11 criteria included in the American College of Rheumatology (ACR) Classification Criteria and/or 4 of the 17 criteria (with at least one of those being clinical and at least one being immunologic) included in the Systemic Lupus International Collaborating Clinics (SLICC) Criteria, at the screening visit.
3. Must have a positive ANA (≥1:160 titer) or positive anti-dsDNA antibody test within 6 months of the screening visit
4. An eGFR of ≥ 30 mL/min/1.73 m2 in the screening period
5. Prior SLE background therapy with at least one non-biologic medication (e.g. immunosuppressant and/or antimalarial), not including corticosteroids, is required for ≥ 12 weeks before the screening visit.
6. SLEDAI-2K ≥6 at the time of screening
7. Participant able and willing to provide written informed consent
8. Must be able and willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria

1. History of any non-systemic lupus erythematosus (non-SLE) disease that required treatment with oral or parenteral corticosteroids for more than a total of 2 weeks within the 12 weeks preceding the screening visit.
2. History of dialysis within 12 months prior to the screening visit or expected need for renal replacement therapy (dialysis or renal transplant) within a six-month period after enrollment.
3. Use of prednisone >0.5 mg/kg/day (or equivalent corticosteroid) in the 4 weeks prior to the screening visit.
4. Any change or addition to a non-biologic immunosuppressant and/ or antimalarial regimen (not including corticosteroids) ≤ 12 weeks prior to the Screening visit.
5. Treatment with an interventional agent within the washout time of 90 days or 5 half-lives prior to Baseline (Day 0), whichever is longer.
6. Receipt of any commercially available biologic agent within the washout period described above prior to Baseline (Day 0).
7. Receipt of prior MSC therapy within the washout time of 52 weeks prior to Baseline (Day 0).
8. Previous treatment with any type of cellular therapy e.g., Tregs or CAR-T cells, with the exception of previous MSCs.
9. Major surgery within 90 days prior to Baseline (Day 0) or major surgery planned during the study period
10. Confirmed positive test for active hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or tuberculosis (TB).
11. Any active infection that has not been adequately treated or completely resolved prior to Baseline (Day 0).
12. History of cancer, apart from adequately treated squamous or basal cell carcinoma of the skin, or cervical carcinoma in situ
13. Pregnant or breast-feeding women and women with intention to become pregnant/to breast-feed during the duration of the trial.
14. Women and men who do not agree to use a medically acceptable form of contraception for the duration of the trial.
15. Any other comorbidity which may render the participant unfit for study participation according to the investigator's judgement.
16. Any other medical condition, which in the opinion of the investigator, may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | day 1 to day 168
  Analysis for the primary endpoint will be descriptive in nature. safety and tolerability will be measured by the number of AEs and SAEs observed. Adverse event incidents will be summarized descriptively. The severity grade of each recorded AE, and their relationship to study treatment will be analyzed. The action taken and outcome will also be analyzed accordingly.

SECONDARY OUTCOMES:
Change from baseline in the SLEDAI 2K following administration | day 1 to day 168
  Total score ranging from 0 to 105.
  Interpretation: Scores are categorized to indicate disease activity:
  0: No activity 1-5: Mild activity 6-10: Moderate activity 11-19: High activity
  ≥20: Very high activity
  Improvement is defined as a decrease in score.
Change from baseline in PROMIS(Patient-Reported Outcomes Measurement Information System) score | day 1 to day 168
  Change from baseline in scores for quality of life, fatigue, pain, and depression as reported by the patient. Scores range from 0 to 100. Higher scores indicate worse symptoms.
Change from baseline in the BILAG-2004 Index score following administration | day 1 to day 168
  Organ involvement is categorized into grades:
  A: Severe active disease B: Moderate active disease C: Stable disease D: Resolved disease E: No involvement
  Improvement is defined as an increase in score.
Efficacy by SRI-4 Responder assessment at Day 168. | day 1 to day 168
  Change from baseline in SRI-4, defined as a ≥4-point reduction in SLEDAI, with no significant worsening in BILAG or PGA. A higher SRI-4 response rate reflects greater clinical improvement.
Change from baseline in prednisone-equivalent corticosteroid doses at each visit performed. | day 1 to day 168.
  Reduction in prednisone-equivalent corticosteroid dose from Day 1 to Day 168.

OTHER OUTCOMES:
Change of pre-treatment versus post-treatment levels of Anti-ENA Antibodies | day 1 to day 168.
  Improvement is defined as a decrease in anti-ENA antibody levels from pre-treatment to post-treatment measurements.
Change of pre-treatment versus post-treatment levels of Anti-dsDNA Antibodies | day 1 to day 168
  Improvement is defined as a reduction in antibody levels.
Change of pre-treatment versus post-treatment levels of Total Serum IgG Levels | day 1 to day 168
  Improvement is defined as a reduction in serum IgG levels.
Change of pre-treatment versus post-treatment results of CBC | day 1 to day 168
  Improvement is defined as any change in values compared to normal range.
Change of pre-treatment versus post-treatment levels of Anti-nucleosome antibodies | day 1 to day 168
  Improvement is defined as a reduction in Anti-nucleosome antibodies levels.
Change of pre-treatment versus post-treatment levels of Erythrocyte sedimentation rate | day 1 to day 168
  Improvement is defined as a reduction in Erythrocyte sedimentation rate.
Change of pre-treatment versus post-treatment levels of CRP | day 1 to day 168
  Improvement is defined as a reduction in CRP levels.
Change of pre-treatment versus post-treatment levels of Cytokines and Chemokines | day 1 to day 168
  Improvement is defined as a reduction in cytokine and chemokine levels.
Change of pre-treatment versus post-treatment Proteinuria measured by protein/creatinine ratio in spot urine | day 1 to day 168
  Improvement is defined as a reduction in protein/creatinine ratio in spot urine
Change of pre-treatment versus post-treatment 24-hour urine protein measured by protein/creatinine ratio in 24-hour urine collection | day 1 to day 168
  Improvement is defined as a reduction in Protein/Creatinine ratio in in 24-hour urine collection
Change of pre-treatment versus post-treatment levels of C3 ; C4 levels | day 1 to day 168
  Improvement is defined as an increase in C3 and/or C4 levels from pre-treatment to post-treatment measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided